CLINICAL TRIAL: NCT06506994
Title: An Open Label, Tolvaptan-controlled Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of Multiple Ascending Dose of HRS-9057 in Heart Failure With Volume Overload
Brief Title: A Study of HRS-9057 in Patients With Heart Failure and Volume Overload
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRS-9057-103
Record Dates: First submitted 2024-06-28; First posted 2024-07-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Heart Failure With Volume Overload
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Intervention Model Description: HRS-9057 injection was compared with Tolvaptan tablets
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group A: HRS-9057/ Tolvaptan (Experimental)
  Interventions: Drug: HRS-9057; Drug: Tolvaptan
- Treatment group B: HRS-9057/ Tolvaptan (Experimental)
  Interventions: Drug: HRS-9057; Drug: Tolvaptan

INTERVENTIONS:
Drug: HRS-9057 — HRS-9057 injection dose 1
  Arms: Treatment group A: HRS-9057/ Tolvaptan
Drug: HRS-9057 — HRS-9057 injection dose 2
  Arms: Treatment group B: HRS-9057/ Tolvaptan
Drug: Tolvaptan — Tolvaptan tablets

SUMMARY:
The study is an open-label, Tolvaptan-controlled Phase I study to evaluate the safety, tolerability, PK/PD profile and efficacy of HRS-9057 in the treatment of heart failure with volume overload. A total of 24 subjects who experience volume overload due to heart failure despite diuretic treatment will be enrolled in the study and receive HRS-9057 injection or Tolvaptan tablets.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18-75 years at the time of signing informed consent.
2. Diagnosed as chronic heart failure at least 1 month prior to screening.
3. Patients with CHF in whom lower limb edema, pulmonary congestion, jugular venous distension or hepatomegaly due to volume overload is present despite diuretics treatment.

Exclusion Criteria:

1. Medical history of myocardial infarction, acute decompensated heart failure, stroke, or transient ischemic attack within 30 days prior to or at screening;
2. Hypovolemic hyponatremia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-10-29 (Actual); Study Completion 2025-10-29 (Actual)

PRIMARY OUTCOMES:
The incidence and severity of any adverse events (AEs) | baseline up to Day 14

SECONDARY OUTCOMES:
Tmax for HRS-9057 | Predose on Day 1 through Day 6
Cmax for HRS-9057 | Predose on Day 1 through Day 6
Daily urine volume | Predose on Day 1 through Day 7
Daily fluid balance | Predose on Day 1 through Day 7
  Daily fluid balance is calculated by subtracting daily urine volume from daily fluid intake.
Serum sodium concentration | Predose on Day 1 through Day 6
Serum osmolality | Predose on Day 1 through Day 6
Urine osmolality | Predose on Day 1 through Day 7
Body weight | baseline to Day 8
Lower limb edema change from baseline | baseline to Day 8
  The severity of edema in the subject's tibial border or dorsum of the foot will be assessed in the sitting position using a 4-point scale (0-absent, 1-mild, 2-moderate and 3-severe) by the investigator. The percentage of subjects in whom the lower limb edema was improved or worsening at Day 8 will be evaluated.
Jugular venous distension change from baseline | baseline to Day 8
  Whether or not the subject has jugular venous distension will be documented. If distension is observed, the vertical height (in centimeters) from the sternal angle to the highest point of pulsation of the internal jugular vein will be documented and the change from baseline to Day 8 will be evaluated.
Pulmonary congestion change from baseline | baseline to Day 8
  The investigator will perform chest X-ray at baseline and Day 8 to assess the severity of pulmonary congestion using a 4-point scale (0-absent, 1-mild, 2-moderate and 3-severe). The percentage of subjects in whom pulmonary congestion was improved or worsening at Day 8 will be evaluated.
New York Heart Association (NYHA) classification change from baseline | baseline to Day 8

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided